CLINICAL TRIAL: NCT00363753
Title: Pilot Study of Continuing Aspirin Versus Switching to Clopidogrel After Stroke or Transient Ischemic Attack
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSD IRB #060452
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Transient Ischemic Attack; Stroke; Aspirin; Clopidogrel
Keywords: Transient ischemic attack; Stroke; Aspirin; Clopidogrel
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

INTERVENTIONS:
Drug: aspirin versus clopidogrel

SUMMARY:
Pilot study of continuing aspirin versus switching to clopidogrel after stroke or transient ischemic attack.

DETAILED DESCRIPTION:
Pilot study of continuing aspirin versus switching to clopidogrel after stroke or transient ischemic attack.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Stroke or transient ischemic attack (TIA) while taking aspirin within one week of consent.
* Women of child-bearing potential will be included only if there is a negative pregnancy test and they agree to birth control during the treatment period.

Exclusion Criteria:

* Any medical indication for a specific antiplatelet agent (aspirin, clopidogrel, ticlopidine, aggrenox), or an indication for a combination of antiplatelet agents.
* Any medical indication for anticoagulation, except subcutaneous heparin for deep vein thrombosis prophylaxis.
* Allergy to aspirin or clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Study Completion 2007-03 (Estimated)

PRIMARY OUTCOMES:
mRS at three months.

SECONDARY OUTCOMES:
Incidence of stroke at three months, bleeding events.

CONTACTS AND LOCATIONS:
Overall Officials: Matt B Jensen, MD, Principal Investigator — UCSD Stroke Center
Locations (2):
- United States (2):
  - UCSD Hillcrest, San Diego, California
  - UCSD, San Diego, California